CLINICAL TRIAL: NCT01583738
Title: Effect of V0251 in Acute Vertigo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V0251 IV 202 4A; 2011-003412-23 (EudraCT Number)
Record Dates: First submitted 2012-04-11; First posted 2012-04-24 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Acute Vertigo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- V0251 (Experimental)
  Interventions: Drug: V0251
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: V0251 — single dose
  Arms: V0251
Drug: placebo — single dose
  Arms: Placebo

SUMMARY:
Assessment of efficacy and tolerance of a new anti-dizziness drug in acute vertigo.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Age 18 to 70 years
* Acute vertigo attack due to vestibular disorder

Exclusion Criteria:

* Signs of brain, brainstem and/or cerebellar dysfunction
* Concomitant central neurological disorder
* Psychogenic vertigo
* Use of ototoxic drugs causing vertigo or dizziness within the last month
* Use of anti-dizziness medications from the onset of symptoms, except if the dosage had been stable for at least 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
"Vertigo Symptoms Score" (VSS) rated by patient using VAS | 30 min

SECONDARY OUTCOMES:
"Concomitant and Vegetative Symptoms Score" (CVSS) rated by patients using VAS | 30 min, 2 hours and 4 hours post dose
Number of patients with Adverse Events as a measure of safety and tolerability | 30 min, 2 hours and 4 hours post dose

CONTACTS AND LOCATIONS:
Locations (40):
- Czechia (7):
  - Fakultni Nemocnice Hradec Králové, Hradec Králové
  - Regional Hospital Kladno, Kladno
  - Faculty Hospital Ostrava, Ostrava
  - Faculty Hospital Královské Vinohrady, Prague
  - Faculty Hospital Motol, Prague
  - Thomayer's Teaching Hospital, Prague
  - Strepomrauska Nemocaicni a. S., Prostějov
- France (5):
  - CHI Elbeuf-Louviers-Val de Reuil, Elbeuf
  - Hôpital Nord, Marseille
  - CHU de Rouen, Hopital Charles Nicolle, Rouen
  - Hôpital Nord, Saint-Etienne
  - Hopital Purpan, Toulouse
- Germany (9):
  - Universitätsklinikum Aachen, Aachen
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Park - Klinik Weissensee, Berlin
  - Allgemeines Krankenhaus Celle, Celle
  - Universitätsklinikum Essen, Essen
  - Goethe-University, Frankfurt am Main
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - University Hospital Mannheim, Mannheim
  - Universitätsklinikum München, München
- Hungary (9):
  - Semmelweis Egyetem Neurológiai Klinika, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum, Debrecen
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Kaposi Mór Megyei Oktató Kórhaz, Kaposvár
  - Borsod Abaúj Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc
  - Kanizsai Dorottya Kórház, Nagykanizsa
  - Pécsi Tudományegyetem Általános Orvostudományi Kar, Pécs
  - Soproni Erzsébet Oktató Kórház, Sopron
  - Markusovszky County Hospital, Szombathely
- Spain (10):
  - Complejo H.Universitario de Badajoz, Badajoz
  - Hospital de Poniente, El Ejido
  - Hospital Universitario de Getafe, Getafe -Madrid
  - Hospital Comarcal San Agustin, Linares
  - Hospital Gregorio Marañón, Madrid
  - Clinica Universitaria de Navarra, Pamplona
  - Complejo Hospitalario de Pontevedra- Montecelo, Pontevedra
  - H. Clínico de Salamanca, Salamanca
  - Hospital Clinico Universitario, Santiago de Compostela
  - Hospital Universitario La Fe, Valencia